CLINICAL TRIAL: NCT04667143
Title: A Multicenter, Randomized, Double-Blind, Parallel Group, Phase 3 Trial to Evaluate the Safety and Efficacy of Retagliptin Plus Henagliflozein Added to Metformin Compared to Retagliptin or Henagliflozein in Combination With Metformin in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin Alone
Brief Title: Dual Add-on Therapy in Type 2 Diabetes Poorly Controlled With Metformin Monotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR3824-SP2086-MET-301
Record Dates: First submitted 2020-12-09; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Retagliptin 100 mg, Henagliflozein 10 mg, plus metformin XR (Experimental)
  Interventions: Drug: Retagliptin, Henagliflozein, metformin XR
- Retagliptin 100 mg, Henagliflozein 5 mg, plus metformin XR (Experimental)
  Interventions: Drug: Retagliptin, Henagliflozein, metformin XR
- Retagliptin placebo, Henagliflozein 10 mg, plus metformin XR (Experimental)
  Interventions: Drug: Retagliptin, Henagliflozein, metformin XR
- Retagliptin placebo, Henagliflozein 5 mg, plus metformin XR (Experimental)
  Interventions: Drug: Retagliptin, Henagliflozein, metformin XR
- Retagliptin 100 mg, Henagliflozein placebo, plus metformin XR (Experimental)
  Interventions: Drug: Retagliptin, Henagliflozein, metformin XR

INTERVENTIONS:
Drug: Retagliptin, Henagliflozein, metformin XR — Retagliptin-DPP4 inhibitor Henagliflozein-SGLT-2 inhibitor Metformin XR

SUMMARY:
2 weeks screening period, 4 weeks run-in period, 24 weeks double-blind treatment period, to evaluate the Safety and Efficacy of Retagliptin Plus Henagliflozein added to Metformin compared to Retagliptin or Henagliflozein in combination with Metformin in Subjects with Type 2 Diabetes who have Inadequate Glycemic Control on Metformin Alone

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, 18-75 years old (both inclusive) at time of screening visit;
2. Subjects with T2DM with inadequate glycemic control defined as central laboratory HbA1c ≥ 7.5 and ≤ 10.5 % at the screening visit;
3. FPG ≤ 15mmol/L at the screening visit;
4. Stable metformin therapy for at least 8 weeks prior to screening at a dose ≥ 1500 mg per day;
5. 19.0<BMI ≤ 40.0 kg/m2 at the screening visit;

Exclusion Criteria:

1. Moderate or severe impairment of renal function [defined as eGFR<60mL/min/1.73 m2 (estimated by MDRD);
2. Uncontrolled hypertension defined as systolic blood pressure (SBP) ≥ 160 mmHg and/or diastolic blood pressure (DBP) ≥ 100 mmHg;
3. Cardiovascular diseases within 6 months of the screening visit;
4. ALT and/or AST > 1.5 x ULN and or Total Bilirubin > 1.2 x ULN;
5. Hemoglobin ≤ 100 g/L;
6. CK (creatine kinase) and CK-MB > 3 x ULN;
7. Malignancy within 5 years of the screening visit (with the exception of treated basal cell or treated squamous cell carcinoma);
8. Administration of any antihyperglycemic therapy, other than metformin,within 2 months prior to screening;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in HbA1c at Week 24 | 24 weeks
  • To compare the mean change from baseline in HbA1c achieved with concurrent addition of Retagliptin Plus Henagliflozein to metformin vs the addition of Retagliptin or Henagliflozein to metformin after 24 weeks of double-blind treatment.